CLINICAL TRIAL: NCT02455804
Title: NIRTRAKS - (NIRxcell TRial for a Post mArKet Study)
Brief Title: NIRTRAKS Post-Market Study (NIRTRAKS)
Acronym: NIRTRAKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV103-02
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: de Novo Stenotic Lesions in Native Coronary Arteries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Other): This is a prospective, post-marketing, non-randomized, multi-center, single-arm clinical study that will be conducted at up to 15 sites in the United States (US). All subjects will be treated with the NIRxcell Stent System and followed at 30 days, 9 months and 1, 2 and 3 years post-index stenting procedure. An unscheduled follow up may be conducted as clinically warranted.
  Interventions: Device: Stenting procedure

INTERVENTIONS:
Device: Stenting procedure — All subjects will be treated with the NIRxcell Stent System and followed at 30 days, 9 months and 1, 2 and 3 years post-index stenting procedure. An unscheduled follow up may be conducted as clinically warranted.

SUMMARY:
This is a prospective, post-marketing, non-randomized, multi-center, single-arm clinical study that will be conducted at up to 15 sites in the United States (US). All subjects will be treated with the NIRxcell Stent System and followed at 30 days, 9 months and 1, 2 and 3 years post-index stenting procedure. An unscheduled follow up may be conducted as clinically warranted.

DETAILED DESCRIPTION:
The main objective of this study is to collect and analyze additional information about the safety and effectiveness of the NIRxcell Stent System in the treatment of de novo stenotic lesions in native coronary arteries in the US population. The primary endpoint will be the rate of target vessel failure (TVF) at 3 years of treatment with the NIRxcell Stent System. This rate will be compared with a performance goal derived from a meta-analysis of coronary stenting with bare metal stents (BMS).

ELIGIBILITY:
Inclusion Criteria:

General

1. Subject is ≥18 years old.
2. Subject is eligible for percutaneous coronary intervention (PCI).
3. Subject is eligible for dual anti-platelet therapy (DAPT) with aspirin plus either clopidogrel, prasugrel or ticagrelor for a minimum of 1 month.
4. Subject understands the nature of the procedure and provides written informed consent prior to the catheterization procedure.
5. Subject is willing to comply with specified follow-up evaluation and can be contacted by telephone.
6. Subject is an acceptable candidate for coronary artery bypass graft (CABG) surgery.
7. Subject has stable angina pectoris (Canadian Cardiovascular Society Classification [CCSC] 1, 2, 3 or 4) or unstable angina pectoris (Braunwald Class 1-3, B-C) or a positive functional ischemia study (e.g. exercise tolerance test [ETT], single-photon emission computerized tomography [SPECT], stress echocardiography or cardiac computerized tomography [CT]).
8. Female subjects of child bearing potential must have a negative pregnancy test within 7 days prior to enrollment in the study.

Angiographic Inclusion Criteria

1. Subject is indicated for elective stenting of a single stenotic lesion in a native coronary artery.
2. Reference vessel ≥2.5 mm and ≤4.0 mm in diameter by visual estimate.
3. Target lesion ≤30 mm in length by visual estimate (the intention should be to cover the whole lesion with 1 stent of adequate length).
4. Target lesion stenosis ≥50% and <100% by visual estimate.

Exclusion Criteria:

General Exclusion Criteria

1. Subject is currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
2. Subject was enrolled in another stent trial within 2 years prior to the index procedure.
3. Any planned elective surgery or percutaneous intervention within 9 months post- procedure.
4. A previous coronary interventional procedure of any kind within 30 days prior to the procedure.
5. The subject requires staged procedure of either the target vessel or any non-target vessel within 9 months post-procedure.
6. The target lesion requires treatment with a device other than percutaneous transluminal coronary angioplasty (PTCA) prior to stent placement (such as, but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.).
7. Previous drug-eluting stent (DES) deployment anywhere in the target vessel.
8. Any previous DES deployment within the past 12 months.
9. Any previous stent placement within 15 mm proximal or distal to the target lesion.
10. Co-morbid condition(s) that could limit the subject's ability to participate in the trial or to comply with follow-up requirements, or impact the scientific integrity of the trial.
11. Concurrent medical condition with a life expectancy of <3 years.
12. Documented left ventricular ejection fraction (LVEF) <25% at the most recent evaluation.
13. Evidence of an acute MI within 72 hours of the intended index procedure.
14. History of cerebrovascular accident or transient ischemic attack within 6 months prior to the index procedure.
15. Leukopenia (leukocytes <3.5 x 109/liter).
16. Neutropenia (absolute neutrophil count <1,000/mm3) ≤ within 7 days prior to enrollment.
17. Thrombocytopenia (platelets <100,000/mm3) pre-procedure (within 7 days prior to enrollment).
18. Active peptic ulcer or active gastrointestinal (GI) bleeding.
19. Subjects who are ineligible for ≥1 month of DAPT because of bleeding diathesis or any other reason.
20. Known hypersensitivity or contraindication to aspirin, thienopyridine, both heparin and bivalirudin, cobalt, nickel, L-605 cobalt chromium alloy or sensitivity to contrast media which cannot be adequately pre-medicated.
21. Serum creatinine level >2.5 mg/dL within 7 days prior to the index procedure.
22. Subject was previously enrolled in the PIONIR Study or the NIRTRAKS Post-Market Study.

Angiographic Exclusion Criteria

1. Unprotected left main coronary artery disease (obstruction >50% in the left main coronary artery that is not protected by ≥1 non-obstructed bypass graft to the left anterior descending [LAD] or left circumflex [LCX] artery or a branch thereof).
2. Target vessel exhibiting multiple lesions with >60% diameter stenosis outside of a range of 5 mm proximal and distal to the target lesion based on visual estimate or on-line quantitative coronary angiography (QCA).
3. Target lesion exhibiting an intraluminal thrombus (occupying >50% of the true lumen diameter) at any time prior to the start of the intervention.
4. Lesion location that is aorto-ostial or within 5 mm of the origin of the LAD or LCX.
5. Target lesion with side branches >2.0 mm in diameter.
6. Target lesion involving a bifurcation (either stenosis of both main vessel and major branch or stenosis of just major branch).
7. Target lesion with severe calcification.
8. Target vessel exhibiting excessive tortuosity that may impede stent delivery and deployment at target lesion.
9. Target lesion that is located in a native vessel distal to an anastomosis with a saphenous vein graft or a left/right internal mammary artery (LIMA/RIMA) bypass.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manesh R Patel, MD, FACC, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 65
Completed | 46
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.06 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 60
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Target Vessel Failure
Description: The primary endpoint in this study was TVF (Target Vessel Failure) defined as a composite of cardiac death, target vessel myocardial infarction (MI), or clinically driven target vessel revascularization (TVR) by percutaneous or surgical methods within 3 years post-procedure.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of TVF
Arm/Group | Single Arm
Number analyzed (Participants) | 61
percentage of TVF | 15 [14.5 to 37.3]

ADVERSE EVENTS:
Time Frame: Adverse events occurring (1) from time of index procedure to 30 days follow-up contact, (2) From 30 days follow up contact to 1 year follow-up contact, (3) From 1 year follow-up contact to 2 years follow-up contact, and (4) From 2 years follow-up contact to 3 years follow-up contact, were recorded.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 40/65
Other Adverse Events (participants affected / at risk) | 58/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=65)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1)
cardiac disorders (Cardiac disorders) | 29 (43)
ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1)
Eye disorders (Eye disorders) | 1 (1)
General disorders and administration site conditions (Gastrointestinal disorders) | 8 (10)
General disorders and administration site conditions (General disorders) | 6 (7)
hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 6 (8)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 5 (8)
Investigations (Investigations) | 1 (1)
metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (3)
musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (4)
neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
nervous system disorders (Nervous system disorders) | 1 (1)
psychiatric disorders (Product Issues) | 1 (1)
renal and urinary disorders (Renal and urinary disorders) | 5 (5)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Vascular disorders (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=65)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5 (5)
Cardiac Disorders (Cardiac disorders) | 37 (69)
ear and labyrinth disorders (Eye disorders) | 1 (1)
Eye disorders (Eye disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 12 (17)
General disorders and administration site conditions (General disorders) | 21 (31)
hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 14 (17)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 7 (10)
Investigations (Investigations) | 5 (5)
metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (5)
musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 7 (11)
neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5)
nervous system disorders (Nervous system disorders) | 9 (10)
psychiatric disorders (Psychiatric disorders) | 2 (2)
renal and urinary disorders (Renal and urinary disorders) | 6 (6)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 19 (28)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Vascular disorders (Vascular disorders) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-03-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT02455804/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT02455804/SAP_001.pdf